CLINICAL TRIAL: NCT03077763
Title: The Effects of Free Haemoglobin NO-blockade on Nitrite Forearm Vessel Dilatation Under Normoxia and Hypoxia in Healthy Volunteers
Brief Title: The Haem and Nitrite Study - The Effects of Haemoglobin NO-blockade on Nitrite-induced Forearm Vessel Dilatation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 206995
Record Dates: First submitted 2016-09-20; First posted 2017-03-13 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
Keywords: nitrite; haemoglobin; normoxia; hypoxia; vasodilatation; blood
MeSH Terms: conditions — Hypoxia; Aneurysm | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normoxia and Nitrite (3umol/min-1) (Active Comparator): Sodium nitrite stock solution: 100umol/10ml, prepared to concentration according to oxygen sequence. Normoxia (3umol/min-1).
  Interventions: Drug: Sodium Nitrite
- Hypoxia and Nitrite (1umol/min-1) (Active Comparator): This will be repeated as per the normoxia cohort, but at a reduced dose of sodium nitrite (1umol/min-1 for 30 minutes) and the volunteers will be asked to breathe 12% oxygen/88% nitrogen for 1-5 minutes before Plethysmography is performed (to get the volunteer to an oxygen saturation of 83-88% peripherally).
  Interventions: Drug: Sodium Nitrite

INTERVENTIONS:
Drug: Sodium Nitrite

SUMMARY:
The study is a pharmacodynamic random order cross-over trial investigating the physiological effects of intra-arterial infusion of nitrite following a haemolysed autologous blood transfusion.

DETAILED DESCRIPTION:
This is a healthy volunteer study.

Following entry into this cross-over trial, participants will be randomized to undergo experiments under either normoxic followed by hypoxic conditions, or hypoxic followed by normoxic conditions.

Subjects will donate whole blood as an autologous unit at a preselected NHSBT donation site. The unit will transported back to the NNUH blood bank after a minimum of 30 days (maximum 35 days) after donation.

Volunteers will be tested for baseline bloods. Volunteers will be randomised to normoxia or hypoxia. The will then undergo a nitrite infusion, followed by an autologous whole blood transfusion and a second nitrite infusion (which will co-infuse at the end of the transfusion). During the protocol, the participants will undergo repeated FBFR measurements using strain-gauge plethysmography.

After a minimum of 12 weeks rest period after their initial donation, participants will cross-over to the opposite oxygen condition (as per initial randomization) and the above protocol will be repeated. All interventions will be performed by fully trained and competent medical staff.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged greater than or equal to 18 years
2. If between 18-20 years of age, calculate total blood volume should be more than >3.5L (http://www.blood.co.uk/giving-blood/who-can-give-blood/)
3. Body weight > 50kg weight (8 stone 12lbs)
4. Not known to have any significant past medical history and not having regular follow up (Check Donor Selection Guidelines (http://www.transfusionguidelines.org.uk/)
5. Willing to provide blood donation and receive autologous blood transfusion
6. After assessment for eligibility pass all blood donor eligibility criteria
7. Able to provide informed consent
8. Should inform overseas travel plan during study period (Check Geographical Disease Risk Index on http://www.transfusionguidelines.org.uk/dsg/gdri) e.g. unable to donate blood for 6 months if travel in a malaria endemic country. Similar guidelines for West Nile virus and T. Cruzi endemic countries.

Exclusion Criteria:

1. Significant medical, surgical or psychiatric disease that in the opinion of the Clinical Research Fellow would affect subject safety or significantly impact his/her ability to comply with follow-up. This would include any known clotting disorders.
2. Known allergy or intolerance to Nitrites
3. Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
4. Female subjects must be of non-childbearing potential, defined as follows: postmenopausal females who have had at least 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhoea with serum FSH>40mIU/ml or females who have had a hysterectomy, bilateral salpingectomy or bilateral oophorectomy at least 6 weeks prior to enrolment
5. Receipt of an investigational drug or biological agent within the 4 weeks prior to study entry or 5 times the drug half-life, whichever is the longer
6. Predisposed to acute on chronic limb ischemia evident from a history of claudication or known peripheral arterial disease.
7. No past history of significant adverse events post blood donation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in FBFR during intra-brachial nitrite and haemolysed blood co-infusion in normoxia vs hypoxia. | Up to 18 months

SECONDARY OUTCOMES:
Change in FBFR during haemolysed blood infusion vs baseline | Up to 18 months
Change in FBFR during nitrite infusion in normoxia vs nitrite infusion in hypoxia | Up to 18 months
Change in FBFR during nitrite infusion in normoxia vs baseline | Up to 18 months
Change in FBFR during nitrite infusion in hypoxia vs baseline | Up to 18 months
Blood analysis (cell free haemoglobin, nitrate, nitrite and nitroso species levels) | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Frenneaux, FRCP, FESC, Principal Investigator — Dean of Medicine, Norwich Medical School, The University of East Anglia, UK
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No